CLINICAL TRIAL: NCT01685307
Title: Impact of Cooking Process on Meat Protein Digestion and Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Manager of the HNRC, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRONUTRIAL
Record Dates: First submitted 2012-03-21; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Physiology; Digestive Tract; Heating Process
Keywords: ileal digestibility; metabolism; stable isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intense cooking process (Experimental): Test meal: 150g of beef cooked at intense temperature. Beef proteins are intrinsically labelled with 15 N protein
  Interventions: Dietary Supplement: Test meal
- mild cooking process (Experimental): Test meal: 150 g of beef cooked at moderate intensity. Beef proteins are intrinsically labeled with 15N.
  Interventions: Dietary Supplement: Test meal

INTERVENTIONS:
Dietary Supplement: Test meal — test meal is 150 g of beef cooked either at moderate or high intensity. Proteins are intrinsically labelled with 15N.

SUMMARY:
Few is known on meat protein digestibility in humans and the impact of cooking process, while excessive intake of processed meat has been suggested to increase the risk of colorectal cancer.

This study aims to measure in vivo in humans the real digestibility of beef meat proteins depending 2 cooking processes, using ileal tubes and stable isotopes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI between 18 an 27
* Age between 18 and 45 years

Exclusion Criteria:

* Gastrointestinal or liver pathology
* Diabetes
* Pregnancy
* Vegetarian

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
protein digestibility | single measure
  From ileal recovery of the ingested tracer during 8 h after the meal

SECONDARY OUTCOMES:
nitrogen metabolism | single measure
  Distribution of dietary nitrogen throug metabolic pools

CONTACTS AND LOCATIONS:
Overall Officials: Claire Gaudichon, PhD, Study Director — INRA AgroParisTech
Locations (1):
- Centre de Recherche sur volontaires, Bobigny, France

REFERENCES:
- [Derived] Oberli M, Marsset-Baglieri A, Airinei G, Sante-Lhoutellier V, Khodorova N, Remond D, Foucault-Simonin A, Piedcoq J, Tome D, Fromentin G, Benamouzig R, Gaudichon C. High True Ileal Digestibility but Not Postprandial Utilization of Nitrogen from Bovine Meat Protein in Humans Is Moderately Decreased by High-Temperature, Long-Duration Cooking. J Nutr. 2015 Oct;145(10):2221-8. doi: 10.3945/jn.115.216838. Epub 2015 Aug 19. PMID 26290008